CLINICAL TRIAL: NCT01925092
Title: An Open-label Study of the Safety, Pharmacokinetics and Pharmacodynamics of Mifepristone in Children With Refractory Cushing's Disease
Brief Title: Mifepristone in Children With Refractory Cushing's Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Corcept Therapeutics (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-CH-0170; 02811-12 (Other: NICHD)
Record Dates: First submitted 2013-08-08; First posted 2013-08-19 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Cushing's Disease
Keywords: Cushing's disease; Mifepristone; Cushing's syndrome; Pharmacokinetic-pharmacodynamic; Child/pediatric population; Safety-efficacy
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; Cushing Syndrome | interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mifepristone (Experimental): Daily doses of mifepristone over 84 days.
  Interventions: Drug: mifepristone

INTERVENTIONS:
Drug: mifepristone — tablets
  Other Names: Korlym

SUMMARY:
Study objectives are to obtain safety, pharmacokinetic, and pharmacodynamic data on the effect of mifepristone on glucose metabolism, body weight and the growth-hormone-IGF in children with refractory Cushing's disease.

DETAILED DESCRIPTION:
The study is being done to examine the effects of a medication called mifepristone in children with Cushing's disease. Since a child's body may absorb and use mifepristone in a different way than adults, it is important to have information about the amount of mifepristone to give children and what will happen to it. Mifepristone has been FDA approved for use only in adults with Cushing's syndrome, and it is important to learn if mifepristone improves the symptoms and signs of Cushing's disease in children. The study is limited to children with Cushing's syndrome due to a pituitary tumor (Cushing's disease) and will not enroll children with Cushing's syndrome due to other causes. The study will investigate how children's bodies absorb and process mifepristone, how it works in children and what effect it has on the use of sugar in the body, on the child's weight and on growth hormone. An important part of the study is to evaluate the side effects of mifepristone in children.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 6-17 years at informed consent
* Active Cushing's disease as demonstrated by the following:
* 24 hour Urinary Free Cortisol greater than the upper limit of normal for age on two urine collections during screening and
* midnight serum cortisol >4.4 mcg/dL (mean of two determinations on a single day at 2330 and 2400 during screening)
* Previous trans-sphenoidal surgery (TSS) for ACTH secreting pituitary tumor at least 3 months prior to screening
* Increased body weight defined by BMI Z-score of 1.5 or above
* Able to provide consent/assent
* Able to swallow study drug tablets (not crushed or split)
* Willing to use non-hormonal method of contraception in patients of reproductive potential
* Primary health care provider in home location

Exclusion Criteria:

* Hypercortisolism not due to Cushing's disease.
* Type 1 diabetes mellitus
* HbA1c ≥9.5% at Screening
* Body weight <25 kg
* Use of certain medications that are CYP3A substrates with narrow therapeutic ranges, such as simvastatin, lovastatin, cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus, and tacrolimus during the 4 weeks prior to starting study drug. Use of these medications is also prohibited until 2 weeks after end of dosing.
* Use of certain medications that are strong CYP3A inhibitors such as itraconazole, nefazodone, ritonavir, nelfinavir, indinavir, atazanavir, amprenavir, fosamprenavir, boceprevir, clarithromycin, conivaptan, lopinavir, mibefradil, posaconazole, saquinavir, telaprevir, telithromycin, and voriconazole during the 2 weeks prior to starting study drug. Use of these medications is also prohibited until 2 weeks after end of dosing. Grapefruit and grapefruit juice, as well as grapefruit-related fruits and their juice (e.g. Seville oranges, pomelos), are prohibited during this time frame.
* Use of certain medications that are strong inducers of CYP3A such as rifampin, rifabutin, rifapentine, phenobarbital, phenytoin, carbamazepine, St. John's wort during the 2 weeks prior to starting study drug. Use of these medications is also prohibited until 2 weeks after end of dosing.
* Use of medications used to treat hypercortisolism from the duration indicated below prior to Day 1. Use of the medications is also prohibited until after the end of study 4 week follow up visit.
* steroidogenesis inhibitors such as ketoconazole, metyrapone: 4 weeks
* cabergoline, bromocriptine, somatostatin analogs such as octreotide, lanreotide, pasireotide long acting formulations: 8 weeks (immediate release formulations: 2 weeks)
* mitotane: 8 weeks
* Use of systemic glucocorticoid medications beginning 1 month prior to screening or anticipated use of these medications except for the treatment of adrenal insufficiency. Use of glucocorticoid medications is prohibited during the study until after the end of study 4 week study visit.
* Inflammatory, rheumatological, proliferative or other disorder(s) that would be anticipated to worsen with glucocorticoid blockade (e.g. inflammatory bowel disease, rheumatoid arthritis, psoriasis, etc.).
* Uncontrolled hypo- or hyperthyroidism.
* Uncorrected hypokalemia (<3.5 mEq/L). The screening period may be used to correct hypokalemia prior to starting study drug. Use of potassium and/or mineralocorticoid antagonists is permitted during the study.
* QTc ≥450 msec on Screening electrocardiogram
* Unexplained vaginal bleeding in females and/or any history of endometrial pathology.
* Positive pregnancy test in females.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | collected during the12 week study and 4 week follow-up period; up to 16 weeks total.
  Patients who have received at least 1 dose of mifepristone will be included in the safety evaluations.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- See also: An Open-Label Study of The Safety, Pharmacokinetics and Pharmacodynamics of Mifepristone in Children With Refractory Cushing's Disease — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-CH-0170.html